CLINICAL TRIAL: NCT06471218
Title: Evaluation of the Efficacy and Safety of Multiple Subcutaneous Injections of SHR-1918 in Patients With Hyperlipidemia in Poor Control: a Multicenter, Randomized, Double-blind, Placebo-controlled Phase II Clinical Trials
Brief Title: Efficacy and Safety of SHR-1918 in Patients With Hyperlipidemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing Suncadia Pharmaceuticals Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR-1918-203
Record Dates: First submitted 2024-06-18; First posted 2024-06-24 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Hyperlipidemia
MeSH Terms: conditions — Hyperlipidemias

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment A:SHR-1918/SHR-1918 Placebo (Experimental)
  Interventions: Drug: SHR-1918; SHR-1918 Placebo
- Treatment B:SHR-1918/SHR-1918 Placebo (Experimental)
  Interventions: Drug: SHR-1918; SHR-1918 Placebo

INTERVENTIONS:
Drug: SHR-1918; SHR-1918 Placebo — SHR-1918/SHR-1918 Placebo,two administration

SUMMARY:
Evaluation of the efficacy and safety of multiple subcutaneous injections of SHR-1918 in patients with hyperlipidemia in poor control: a multicenter, randomized, double-blind, placebo-controlled phase II clinical trials

ELIGIBILITY:
Inclusion Criteria:

1. On the day of signing the informed consent form, the age must be ≥ 18 years old and ≤ 75 years old, both men and women are eligible;
2. Screen spatiotemporal abdominal LDL-C for ASCVD risk assessment, meeting the relevant conditions;
3. TG≤5.6mmol/L.

Exclusion Criteria:

1. Alanine aminotransferase (ALT), aspartate aminotransferase (AST), or gamma glutamyltransferase (GGT) exceeding 3 times the ULN, or total bilirubin exceeding 2 times the ULN;
2. Human immunodeficiency virus antibody (HIV Ab), hepatitis C virus antibody (HCV Ab), any of the above test results are positive; Hepatitis B virus surface antigen (HBsAg) positive and HBV-DNA ≥ 1000 copies/ml (or ≥ 200 IU/ml, if the lower limit of the detection value is higher than 1000 copies/ml or 200 IU/ml, HBV-DNA ≥ the lower limit of the detection value);
3. Creatine kinase (CK) exceeds 3 times the upper limit of normal value (ULN);
4. Thyroid stimulating hormone (TSH) is below the lower limit of normal (LLN) or exceeds 1.5 times the upper limit of normal (ULN);
5. Glomerular filtration rate (eGFR)<30 ml/min/1.73m2 (calculated using the MDRD formula, eGFR (mL/min/1.73m2)=175 x (serum creatinine/88.4) -1.234 x age -0.179 x (0.79 females), where serum creatinine units are μ mol/L).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2024-07-02 (Actual); Primary Completion 2025-05-16 (Actual); Study Completion 2025-05-16 (Actual)

PRIMARY OUTCOMES:
Percent change in calculated LDL-C from baseline to week 24 | from baseline to week 24

SECONDARY OUTCOMES:
Percent change in calculated TG from baseline to week 24 | from baseline to week 24

CONTACTS AND LOCATIONS:
Locations (1):
- Meizhou People's Hospital, Meizhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided